CLINICAL TRIAL: NCT06815094
Title: Role of Erector Spinae Plane Block Versus Caudal Epidural Block in Alleviating Intra- & Post-operative Pain in Pediatric Patients Undergoing Lower Limb Cancer Surgeries
Brief Title: Erector Spinae Plane Block Versus Caudal Epidural Analgesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2211-301-044
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2022-11

CONDITIONS: Surgical Pain
MeSH Terms: interventions — Parapsychology

STUDY DESIGN:
Intervention Model Description: randomized parallel group clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of patients received Caudal Epidural Analgesia (Active Comparator): Pediatric patients aged 8 to 15 years of age undergoing unilateral lower limb cancer surgery are recruited from National Cancer Institute & randomly allocated to this group.
  Interventions: Procedure: Regional analgesia either CEA or ESP
- Group of patients received Erector Spinae Plane block (Active Comparator): Pediatric patients aged 8 to 15 years of age undergoing unilateral lower limb cancer surgery are recruited from National Cancer Institute & randomly allocated to this group.
  Interventions: Procedure: Regional analgesia either CEA or ESP

INTERVENTIONS:
Procedure: Regional analgesia either CEA or ESP — Ultrasound guided local anesthetic injection in the course of the conducting nerve to decrease pain transmission.

SUMMARY:
The goal of this clinical trial is to compare the analgesic effect and safety of erector spinae plane block vs caudal epidural block in paediatric population undergoing lower limb cancer surgery. The main questions it aims to answer are:

* Which of them has a superior analgesic effect.
* which of them is more safe and has less complication rate. Participants or their guardians should agree to share in the study (after full explanation of risks and benefits) to receive one of the previously mentioned regional blocks in conjunction with the classic balanced general anaesthesia.

DETAILED DESCRIPTION:
This randomized parallel group clinical trial was carried out on 32 paediatric patients aged from 8 to 15 years old, both sexes, belonging to American Society of Anaesthesiologists II physical status, cancer patient receiving chemotherapy undergoing unilateral lower limb cancer surgery. Patients were divided into two equal groups: Group A: patients received selective unilateral ESPB and group B: patients received CEB. Both in conjunction with general anaesthesia. The primary outcomes were determining the postoperative time of first rescue analgesia and assessment of total postoperative morphine consumption using erector spinae block compared to CEB in the first 12 hours after surgery. The secondary outcomes were assessments of the pain severity intra- and post-operative parallel with recording any complication regarding drugs or procedures.

ELIGIBILITY:
Inclusion Criteria:

* ASA ( American Society of Anaesthesiologists) II (Cancer patient receiving chemotherapy).
* 8 - 15 years of age.
* Planned to undergo unilateral lower limb cancer surgery.

Exclusion Criteria:

* Patients with coagulopathy with INR (International Normalization Ratio) > 1.6 (e.g.: haemophilia, fibrinogen abnormalities and deficiency with concentration < 60 %).
* History of allergy to local anaesthetics or any of the additives.
* Patients refused to be included in the study or their guardians.
* CNS (Central Nervous System) pathology.
* Unstable cardiovascular disease.
* Local or systemic infection.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Determining the actual postoperative time of need for the first rescue analgesia | Immediately and up to the first 12 hours post-operatively.
  Compare the actual postoperative time of need for the first rescue analgesia by the Numerical Rating Score in all cases in both groups when it is equal to or more than 4.
Assessment of total postoperative morphine consumption using erector spinae block compared to CEB in the first 12 hours after surgery. | Immediately and up to the first 12 hours post-operatively.
  Calculation of total postoperative morphine consumption in both groups.

SECONDARY OUTCOMES:
Assessments of the pain severity intra- and post-operatively. | Intraoperatively and up to 12 hours postoperatively.
  Using Numerical Rating Score for postoperative pain assessment and vital data with fentanyl consumption for intraoperative pain assessment.
Recording any complication regarding drugs or procedures. | Intraoperatively and up to 12 hours postoperatively.
  for example hypotension or local anaesthetic toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Atef Badran, MD, Study Director — National cancer institute - Cairo university
Locations (1):
- National Cancer Institute, Cairo, ELkhalig, Egypt

IPD SHARING:
Plan to Share IPD: No